CLINICAL TRIAL: NCT02442674
Title: A Pilot Phase 3b,Multicenter,Randomized,Double-blind,Placebo-controlled Trial of the Safety,Efficacy,and Pharmacokinetics of Titrated Oral SAMSCA®(Tolvaptan) in Children and Adolescent Subjects With Euvolemic or Hypervolemic Hyponatremia
Brief Title: A Trial of Tolvaptan in Children and Adolescent Subjects With Euvolemic and Hypervolemic Hyponatremia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial withdrawn due to inability to meet the trial objectives (Pilot).
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 156-13-207
Record Dates: First submitted 2015-05-08; First posted 2015-05-13 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Hyponatremia
Keywords: Hyponatremia; Euvolemic; Hypervolemic; Serum sodium; Dilutional hyponatremia; Electrolyte abnormality; Electrolyte imbalance; Metabolic disease; Water-Electrolyte Imbalance
MeSH Terms: conditions — Hyponatremia; Metabolic Diseases; Water-Electrolyte Imbalance | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolvaptan (Active Comparator): Tolvaptan (3.75 mg, 7.5 mg, 15 mg, 30 mg, 60 mg dose daily depending on age and weight)
  Interventions: Drug: Tolvaptan
- Placebo (Placebo Comparator): Placebo tablet matching active drug
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan 3.75-, 7.5-, 15-, and 30-mg Tablets.
  Dosage: Depending on age, weight and serum sodium response:
  Tablet (3.75 mg - 60 mg daily) Frequency: Once daily Duration: 30 (+2) days
  Other Names: SAMSCA
  Arms: Tolvaptan
Other: Placebo — Placebo tablet matching active drug
  Arms: Placebo

SUMMARY:
The purpose of this trial is to demonstrate that tolvaptan effectively and safely increases and maintains serum sodium concentrations in children and adolescent subjects with euvolemic or hypervolemic hyponatremia.

DETAILED DESCRIPTION:
The purpose of the study is to also assess tolvaptan's pharmacokinetics (PK) and its effect on fluid balance in children and adolescent subjects with euvolemic or hypervolemic hyponatremia. Subjects who are diagnosed with euvolemic or hypervolemic hyponatremia (serum sodium < 130 mEq/L [mmol/L]) that persists despite initial standard background therapy (eg, including fluid restriction) are eligible to be screened for participation in this trial. Subjects who demonstrate prior resistance to vasopressin antagonist therapy will be excluded. All potential subjects must be deemed by the investigator as likely to benefit from a therapy that raises serum sodium levels.

Subjects will be required to be in a hospital setting during initiation or titration of tolvaptan. Overall, in this trial, subjects will undergo treatment with tolvaptan or placebo for 30 (+2) days and a post-last dose follow-up phase of 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥ 4 years of age (or per local Health Authority age restriction) to < 18 years old and ≥ 10kg
2. Subjects hospitalized with euvolemic or hypervolemic hyponatremia resistant to initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist) and who are deemed by the investigator as likely to benefit from a therapy that raises serum sodium levels
3. Persistent euvolemic or hypervolemic hyponatremia defined as being documented as present for at least 48 hours, evidenced by at least 2 serum sodium assessments < 130 mmol/L drawn at least 12 hours apart (these values can be documented using historical values previously obtained per standard of care); a third (STAT) serum sodium assessment < 130 mmol/L, which will serve as the baseline value for efficacy endpoints, is to be obtained within 2-4 hours prior to the final trial qualification and the first dose of IMP
4. Ability to swallow tablets
5. Ability to maintain adequate fluid intake whether orally or via IV support with adequate monitoring
6. Ability to comply with all requirements of the trial
7. Trial-specific written informed consent/assent obtained from a parent/legal guardian or legally acceptable representative, as applicable per age of subject or local laws, prior to the initiation of any protocol required procedures. In addition, the subject as required by local laws must provide informed assent at Screening and must be able to understand that he or she can withdraw from the trial at any time.

   All informed consent/assent procedures must be in accordance with the trial center's IRB/IEC and local regulatory requirements
8. Ability to commit to remain fully abstinent (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] or withdrawal are not acceptable methods of contraception) or practice double-barrier birth control during the trial and for 30 days following the last dose of IMP for sexually active females of childbearing potential

Exclusion Criteria:

1. Has evidence of hypovolemia or intravascular volume depletion (eg, hypotension, clinical evidence of volume depletion, response to saline challenge); if the subject has systolic blood pressure or heart rate outside of the normal range for that age volume status should be specifically clinically assessed to rule out volume depletion
2. Has serum sodium < 120 mmol/L, with or without associated neurologic impairment (ie, symptoms such as apathy, confusion, or seizures)
3. Subjects ≤ 50 kg taking potent CYP3A4 inhibitors or subjects < 20 kg taking moderate CYP3A4 inhibitors within 72 hours prior to dosing
4. Lacks free access to water (inability to respond to thirst) or without ICU-level fluid monitoring and management
5. Has a history or current diagnosis of nephrotic syndrome
6. Has transient hyponatremia likely to resolve (eg, head trauma or post-operative state)
7. Has hyperkalemia defined as serum potassium above the ULN for the appropriate pediatric age range
8. Has eGFR < 30 mL/min/1.73 m2 calculated by the following equation:

   eGFR (mL/min/1.73 m2) = 0.413 x height (cm)/serum creatinine (mg/dL)
9. Has AKI from recent medical history defined as:

   * Increase in serum creatinine by ≥ 0.3 mg/dL (≥ 26.5 µmol/L) within 48 hours; or
   * Increase in serum creatinine to ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or
   * Urine volume < 0.5 mL/kg/h for 6 hours
10. Has severe or acute neurological symptoms requiring other intervention (eg, hyperemesis, obtundation, seizures)
11. Has had treatment for hyponatremia with:

    * Hypertonic saline (including normal saline challenge) within 8 hours of qualifying serum sodium assessments;
    * Urea, lithium, demeclocycline, conivaptan, or tolvaptan within 4 days of qualifying serum sodium assessments;
    * Other treatment for the purpose of increasing serum sodium concurrent with dosing of IMP
12. Has anuria or urinary outflow obstruction, unless the subject is, or can be, catheterized during the trial
13. Has a history of drug or medication abuse within 3 months prior to Screening or current alcohol abuse
14. Has a history of hypersensitivity and/or idiosyncratic reaction to benzazepine or benzazepine derivatives (such as benazepril)
15. Has psychogenic polydipsia (subjects with other psychiatric illness may be included per medical monitor approval)
16. Has uncontrolled diabetes mellitus, defined as fasting glucose > 300 mg/dL (16.7 mmol/L)
17. Has screening liver function values (ALT/AST) > 3 x ULN
18. Has cirrhosis and meets any of the following conditions: a major GI bleed within the past 6 months, evidence of active bleeding (eg, epistaxis, petechiae/purpura, hematuria, or hematochezia), platelet count < 50,000/µL, or use of concomitant medications known to increase bleeding risk
19. Has hyponatremia due to the result of any medication that can safely be withdrawn (eg, thiazide diuretics)
20. Has hyponatremia (eg, hyponatremia in the setting of adrenal insufficiency, untreated hypothyroidism, or hypotonic fluid administration) that is most appropriately corrected by alternative therapies
21. Is currently pregnant or breastfeeding
22. Has any medical condition that, in the opinion of the investigator, could interfere with evaluation of the trial objectives or safety of the subjects.
23. Is deemed unsuitable for trial participation in the opinion of the investigator
24. Participation in another investigational drug trial within the past 30 days, without prior approval from the sponsor medical monitor
25. Subjects < 4 years of age or per local Health Authority age restriction, weight < 10 kg, or who are unable to swallow tablets are excluded until an alternate formulation becomes available

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Change in serum sodium concentration | Daily up to day 4
  The average daily area under the curve (AUC) of change from baseline in serum sodium level up to Day 4 within the double-blind treatment period.

SECONDARY OUTCOMES:
Change of average daily AUC from baseline at each visit in serum sodium level. | Daily up to Day 30
Change from baseline in serum sodium concentration at Day 4. | Day 4
Change from baseline in serum sodium concentration at Day 30. | Daily up to Day 30
Percentage of subjects who require rescue therapy or fluid restriction at any time during the double-blind treatment period. | Daily up to Day 30
Changes from baseline in ALT, AST and Total Bilirubin | Daily up to Day 30
Clinically significant changes in vital signs. | Daily up to Day 30
Incidence of dehydration AEs. | Daily up to Day 30
Tanner staging progression score (at 30 days) | Daily up to Day 30
Percentage of subjects with overly rapid correction in serum sodium ( ≥ 12 mmol/L in 24 hours). | Daily up to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Ann Dandurand, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.